CLINICAL TRIAL: NCT02600104
Title: Clinical Study to Evaluate the Performance of the PicoWayTM Picosecond Fractional Laser for Wrinkles Reduction
Brief Title: Evaluate the Performance of the PicoWayTM Picosecond Fractional Laser for Wrinkles Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF17271
Record Dates: First submitted 2015-10-28; First posted 2015-11-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Unwanted Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): will receive up to four (4) facial treatments in 3-8 weeks interval, with the PicoWayTM device-fractional hand piece 1064nm and/or 532nm according to the study protocol. Subjects will be followed by phone 7 days post first treatment by study staff, and will return for follow-up (FU) visits at the clinic at: 6 weeks and 12 weeks following the last treatment.
  Interventions: Device: PicoWayTM

INTERVENTIONS:
Device: PicoWayTM — The PicoWayTM base unit using a single, free-running, flashlamp-pumped alexandrite laser as a pump source for both the oscillator and the amplifier

SUMMARY:
Prospective clinical study, Up to 100 healthy adult volunteers seeking Treatment of Wrinkles Reduction in the facial area, males or females of 18 to 75 years of age, from up to 5 investigational sites.

DETAILED DESCRIPTION:
This is an open-label, multi-center study. Subjects in this study will receive up to four (4) facial treatments in 3-8 weeks interval, with the PicoWayTM device-fractional hand piece 1064nm and/or 532nm according to the study protocol. Subjects will be followed by phone 7 days post first treatment by study staff, and will return for follow-up (FU) visits at the clinic at: 6 weeks and 12 weeks following the last treatment.

Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 75 years of age
2. Has Fitzpatrick skin type I-VI
3. Subjects seeking treatment for wrinkles reduction and willing to undergo laser treatments for improvement
4. Have mild to moderate bilateral perioral and/or periorbital wrinkles
5. Willing to receive the proposed PicoWayTM fractional treatments and comply with all study (protocol) requirements
6. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications and presentations (subject identity will be masked)
7. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
8. Informed consent process is completed and subject consent is signed

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
2. Hypersensitivity to light exposure
3. Active sun tan in facial area
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
5. Is taking medication(s) for which sunlight is a contraindication
6. Has a history of squamous cell carcinoma or melanoma
7. History of keloid scarring, abnormal wound healing and / or prone to bruising
8. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders
9. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment, e.g., lack of noticeable skin flaking, skin peeling and skin surface roughness.
10. A laser procedure, a peel or has used lightening creams that was performed in the area to be treated with the past six months
11. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
12. Known allergy to lidocaine, tetracaine, Xylocaine or epinephrine
13. Subjects with pigmented lesions that are considered not acceptable by the study investigator or any condition that, in the investigator's opinion, would make it unsafe to treat.
14. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PicoWay for facial wrinkles reduction treatment assessed by blinded evaluators based on Fitzpatrick Classification and Degree of Elastosis. | day 0 up to 9 months
  assessed by blinded evaluators.

SECONDARY OUTCOMES:
Improvement in Fitzpatrick Classification and Degree of Elastosis, as assessed by study investigator | from 3 weeks up to 9 months
  Percentage of subjects with improvement in Fitzpatrick Classification and Degree of Elastosis, as assessed by study investigator
Safety of PicoWay treatment by Adverse events record during all study | day 0 up to 9 months
  assessed by study investigator during all study
Evaluate investigator satisfaction assessed by questionnaire | from 24 weeks up to 36 weeks
  by questionnaire
Evaluate subject satisfaction assessed by questionnaire | from 24 weeks up to 36 weeks
  by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric F Bernstein, M.D., Principal Investigator — Main Line Center for Laser Surgery
Locations (4):
- United States (4):
  - Jerome M. Garden, Chicago, Illinois
  - Arielle N. Kauvar, New York, New York
  - Eric F. Bernstein, Ardmore, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bloom BS, Emer J, Goldberg DJ. Assessment of safety and efficacy of a bipolar fractionated radiofrequency device in the treatment of photodamaged skin. J Cosmet Laser Ther. 2012 Oct;14(5):208-11. doi: 10.3109/14764172.2012.724534. PMID 23016529